CLINICAL TRIAL: NCT05696782
Title: Phase II Pilot Study of Quick Start Durvalumab Following Chemoradiation for Stage III Nonsmall Cell Lung Cancer
Brief Title: Quick Start Durvalumab Following Chemoradiation for Stage III Nonsmall Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00092850; WFBCCC 62422 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Nonsmall Cell Lung Cancer Stage III; Unresectable Non-Small Cell Lung Carcinoma; Nonsmall Cell Lung Cancer, Stage II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Quick Start Durvalumab (Experimental): Standard of care test and procedures for cancer treatments along with Durvalumab treatment at physician's discretion
  Interventions: Drug: Durvalumab; Other: the EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30); Diagnostic Test: COPD Assessment Test (CAT); Diagnostic Test: Modified Medical Research Council (mMRC) dyspnea scale

INTERVENTIONS:
Drug: Durvalumab — Participants will receive Durvalumab 1500 mg intravenously every two weeks for 60 minutes. Each treatment is called a cycle and lasts for four weeks (or 28 days).
Other: the EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) — Participants will be asked to answer all 30 items on the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). This patient-reported outcome measure is designed to measure cancer patients' physical, psychological and social functions. The measure can be completed using a paper form, by verbally providing answers to the study team, or by entering the answers online into REDCap using a computer or mobile device. The total time to complete the questionnaire is approximately 11 minutes (
Diagnostic Test: COPD Assessment Test (CAT) — Participants will be asked to answer all items on the COPD assessment test (8 items) and the patient-reported outcome measures designed to measure respiratory function. The measures can be completed using a paper form, by verbally providing answers to the study team, or by entering the answers online into REDCap using a computer or mobile device. The total time to complete the questionnaire is less than 5 minutes.
Diagnostic Test: Modified Medical Research Council (mMRC) dyspnea scale — Participants will be asked to answer the modified medical research council dyspnea scale (1 item), and the patient-reported outcome measures designed to measure respiratory function. The measures can be completed using a paper form, by verbally providing answers to the study team, or by entering the answers online into REDCap using a computer or mobile device. The total time to complete the questionnaire is less than 5 minutes.

SUMMARY:
This research study aims to determine what effects (good and bad) Durvalumab has on participants and their cancer with a "quick start" of Durvalumab within 14 days of finishing chemotherapy and radiation. The study will also determine the logistic barriers to the quick start of Durvalumab.

DETAILED DESCRIPTION:
Primary Objective: Assess the treatment fidelity for early Durvalumab initiation (i.e., within 14 days after the last day of radiation therapy) following chemoradiation for unresectable Stage II or Stage III nonsmall cell lung cancer.

Secondary Objectives:

* Assess the treatment fidelity for very early Durvalumab initiation (i.e., within seven days after the last day of radiation therapy) following chemoradiation for unresectable Stage II or Stage III nonsmall cell lung cancer.
* Assess barriers to earlier Durvalumab initiation following chemoradiation for unresectable Stage II or Stage III nonsmall cell lung cancer.
* Describe the toxicity of Durvalumab when initiated quickly after chemoradiation for unresectable Stage II or Stage III nonsmall cell lung cancer as compared to historical controls.
* Describe the efficacy of Durvalumab when initiated quickly after chemoradiation for unresectable Stage II or Stage III nonsmall cell lung cancer as compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage II or Stage III nonsmall cell lung cancer confirmed by histologic or cytologic documentation and by clinical assessment. Staging is defined according to the American Joint Committee on Cancer Staging Manual, 8th Edition (2017).
* Unresectable or medically inoperable as determined by the investigator.
* The participant has definitive radiation therapy (e.g., 54 Gy to 66 Gy in 30 to 35 fractions) for lung cancer that is either (a) planned to start within the next 28 days, or (b) currently being administered, or (c) has been completed within the last 14 days.
* Platinum-based chemotherapy for lung cancer that is either (a) planned to start within the next 28 days, (b) currently being administered, or (c) has been completed within the last 14 days. Chemotherapy must be for at least two cycles and be administered either before radiation therapy ("induction" or "sequential") or during radiation therapy ("concurrent").
* Consolidation Durvalumab is planned for nonsmall cell lung cancer after radiation and chemotherapy.
* Eighteen years old or greater.
* ECOG performance status of 0-2.
* Life expectancy of greater than three months.
* Patients with sexual relationships in which either they or their partner may become pregnant must use contraception during the study treatment period.
* Ability to understand and be willing to sign an IRB-approved informed consent document directly or via a legally authorized representative.

Exclusion Criteria:

* Uncontrolled respiratory symptoms (i.e., cough, dyspnea, fevers, chest pain, or an increase from baseline oxygen requirements) that are interfering with activities of daily living.
* Nonsmall cell lung cancer is known to have a tumor with a mutation in EGFR associated with sensitivity to first-line therapy with a tyrosine kinase inhibitor (i.e., Ex19del or L858R). Testing for EGFR mutation must have been attempted for study enrollment. If EGFR testing is inconclusive (e.g., the biopsy's quantity or quality is not sufficient for testing to be performed) and there is low clinical suspicion for the presence of an EGFR mutation as determined by the investigator, then the patient is eligible.
* Prior exposure to an immune checkpoint inhibitor targeting CTLA-4, PD-1, or PD-L1.
* Active autoimmune disease requiring systemic immunosuppression at the time of enrollment.
* History of autoimmune pneumonitis requiring high-dose systemic steroids (equivalent prednisone >20 mg/day for more than one week).
* Uncontrolled intercurrent illness includes ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants to Achieve Fidelity to Early Treatment with Durvalumab - Early Initiation (1-14 days) | 48 weeks
  Fidelity is defined as a dichotomous composite indicator (yes/no) that describes whether the patient received very early (1-7 days) initiation of Durvalumab as per protocol with all four of the following criteria having been met: (i) CT chest obtained after the last day of radiation therapy and before the first infusion of Durvalumab, (ii) first infusion within 14 days of completing radiation therapy, (iii) second and third doses received within 63 days of the first dose, and (iv) all infusions at least 28 days apart.

SECONDARY OUTCOMES:
Number of Participants to Achieve Fidelity to Early Treatment with Durvalumab - Very Early (1-7 days) | Up to 13 months
  Fidelity is defined as a dichotomous composite indicator (yes/no) that describes whether the patient received very early (1-7 days) initiation of Durvalumab as per protocol with all four of the following criteria having been met: (i) CT chest obtained after the last day of radiation therapy and before the first infusion of Durvalumab, (ii) first infusion within 7 days of completing radiation therapy, (iii) second and third doses received within 63 days of the first dose, and (iv) all infusions at least 28 days apart.
Number of Barriers to Initiation of Durvalumab - Very Early (Days 1-7) | Up to 13 months
  Descriptive frequencies of participant survey answers will be examined to conduct qualitative analyses and determine appropriate categories of answers on the free text responses. We will examine barriers/obstacles for everyone in the sample, even those who achieve fidelity; such patients could have experienced delays even if they were still able to achieve fidelity. We will stratify answers/responses by fidelity status.
Number of Barriers to Initiation of Durvalumab - Early (Days 8-14) | Up to 13 months
  Descriptive frequencies of participant survey answers will be examined to conduct qualitative analyses and determine appropriate categories of answers on the free text responses. We will examine barriers/obstacles for everyone in the sample, even those who achieve fidelity; such patients could have experienced delays even if they were still able to achieve fidelity. We will stratify answers/responses by fidelity status.
Number of Participants with All Adverse Events | Up to 13 months after intervention
  Adverse events, serious adverse events and immune-related adverse events will be tabulated by fidelity status (1-7 days vs. 8-14 days vs. neither) using National Cancer Institute Common Terminology Criteria, version 5.0.
Number of Participants Who Have Immune-Mediated Pneumonitis - Early Fidelity (1-14 days) | Within 85 days of intervention (Cycles 1-3)
  Participants with early (1-14 days) fidelity who have immune-mediated early-onset pneumonitis will be estimated and statistically compared in a one-sample test of proportions.
Number of Participants Who Have All-Cause Any Grade Pneumonitis - Early Fidelity (1-14 days) | Within 85 days of intervention (Cycles 1-3)
  Participants with all-cause early-onset pneumonitis among those with early (1-14 days) fidelity and statistically compare it, using a one-sample test of proportions.
Number of Participants to Discontinue Durvalumab Due to Adverse Events | One year
  Participants with early fidelity who discontinue Durvalumab at any point due to an adverse event of any cause and compare it using a one-sample test of proportions.
Overall Survival | One year
  Using Kaplan-Meier life table methods, overall survival is defined as the number of participants alive at 12 months after the first dose of Durvalumab.
Progression-Free Survival | One year
  Using Kaplan-Meier methods, progression-free survival is defined as the number of participants alive and without disease progression as documented by the treating provider at 12 months after the first dose of Durvalumab.
Response Rate | One year
  Best objective response rate (ORR) to Durvalumab is defined by either a complete response (CR) or partial response (PR) as per RECIST 1.1 criteria by investigator assessment and confirmed on at least two sequential imaging studies that are at least four weeks apart.
  * Complete Response (CR): Disappearance of all target lesions.
  * Partial Response (PR): Decrease by ≥ 30% in sum of longest diameter of target lesions.

OTHER OUTCOMES:
Change in Patient-Reported Outcomes Scores (PROs) - European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Version 3 | Baseline to 12 weeks after start of intervention
  The change in PROs scores from baseline to week 12 using paired t-tests and compare mean difference scores to the null hypothesis value of zero change to compare between fidelity status (1-7 days vs. 8-14 days vs. neither). Scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Change in Patient-Reported Outcomes Scores (PROs) - Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) Questionnaire | Baseline to 12 weeks after start of intervention
  The QLQ-LC13 includes questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea and site specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication. The change in PROs scores from baseline to week 12 using paired t-tests and compare mean difference scores to the null hypothesis value of zero change to compare between fidelity status (1-7 days vs. 8-14 days vs. neither). Scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Change in Respiratory Patient Reported Outcomes (PROs) - COPD Assessment Test (CAT) | Baseline to 12 weeks after start of intervention
  The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD). It is designed to measure the impact of COPD on a person's life and how this changes over time. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD. The change in PROs scores using paired t-tests and compare mean difference scores to the null hypothesis value of zero change to compare between fidelity status (1-7 days vs. 8-14 days vs. neither).
Change in Respiratory Patient Reported Outcomes (PROs) - Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline to 12 weeks after start of intervention
  The mMRC (Modified Medical Research Council) Dyspnea Scale is used to assess the degree of baseline functional disability due to dyspnea.The mMRC breathlessness scale ranges from grade 0 to 4 with grade 4 indicating a higher level of respiratory disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lycan, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No